CLINICAL TRIAL: NCT01001130
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Effectiveness of Avamys® Administered in Korean Patients According to the Prescribing Information
Brief Title: Regulatory AVAMYS Nasal Spray PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113596
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: avamys; Allergic Rhinitis; post marketing surveillance; Seasonal Allergic Rhinitis; Perennial Allergic Rhinitis (PAR)
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fluticasone furoate group: Korean patients administered fluticasone furoate according to the Prescription information
  Interventions: Drug: fluticasone furoate group

INTERVENTIONS:
Drug: fluticasone furoate group — patients who are administered fluticasone furoate at least once
  Other Names: according to label and physician's decision

SUMMARY:
Non-interventional, open-label, single group, multicentric post-marketing surveillance to monitor the safety and effectiveness of AVAMYS nasal spray administered in Korean patients according to the prescribing information.

AVAMYS is a registered trademark of the GSK group of companies.

ELIGIBILITY:
All subjects must satisfy the following criteria.

1. Subject who is treated with AVAMYS nasal spray for the first time.
2. Subject who is treated due to symptoms of seasonal and perennial allergic rhinitis in adults and children ≥2 years.
3. Subject who is considered to follow the PMS protocol by an investigator.
4. Subject who is contactable via telephone.
5. Subject who is treated with AVAMYS nasal spray according to its prescribing information.

As considering the characteristic of the observational post marketing surveillance, the exclusion criteria is not strict. All investigators should prescribe AVAMYS nasal spray according to prescribing information which approved in Korea.

All subjects must not satisfy the following criteria.

1. Subject who has hypersensitivity to its ingredients.
2. As corticosteroids can slow the healing of wounds, if a subject who has surgery on his/her nose recently, or has a sore in his/her nose, or if his/her nose has been injured, the subject does not use AVAMYS nasal spray until his/her nose has healed.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated AVAMYS nasal spray at the site
Sampling Method: Probability Sample
Enrollment: 3244 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with an adverse event | 2 weeks
  Number of participants with an adverse event

SECONDARY OUTCOMES:
Number of participants with a serious adverse event | 2 weeks
  Number of participants with a serious adverse event
Number of participants with an unexpected or expected adverse drug reaction | 2 weeks
  Number of participants with an unexpected or expected adverse drug reaction
Effectiveness after AVAMYS nasal spray administration | 2 weeks
  Effectiveness after AVAMYS nasal spray administration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seongnam-si Gyeonggi-do, South Korea